CLINICAL TRIAL: NCT06492785
Title: Use of Hyaluronic Acid-enriched Transfer Medium in Women Undergoing Single Blastocyst Transfer : a Multicenter, Randomized Controlled Trial
Brief Title: Hyaluronic Acid-enriched Transfer Medium in Single Blastocyst Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Collaborators: Jiangxi Maternal and Child Health Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, He Cai, Principal Investigator, Northwest Women's and Children's Hospital, Xi'an, Shaanxi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-127
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Infertility
Keywords: Hyaluronate-enriched medium; live birth; Single blastocyst transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid(EmbryoGlue®) (Experimental): High HA concentrations (0.5 mg/ml)
  Interventions: Biological: High Hyaluronic Acid concentrations (0.5 mg/ml)
- Hyaluronic Acid (G2 medium) (Active Comparator): Low HA concentrations (0.125 mg/ml)
  Interventions: Biological: Low Hyaluronic Acid concentrations (0.125 mg/ml)

INTERVENTIONS:
Biological: High Hyaluronic Acid concentrations (0.5 mg/ml) — Hyaluronic Acid(EmbryoGlue®)
  Arms: Hyaluronic Acid(EmbryoGlue®)
Biological: Low Hyaluronic Acid concentrations (0.125 mg/ml) — Hyaluronic Acid (G2 medium)
  Arms: Hyaluronic Acid (G2 medium)

SUMMARY:
The purpose of this study is to compare the live birth rates of high concentration of Hyaluronic Acid (0.5 mg/ml) transfer medium (EmbryoGlue®) to those containing low Hyaluronic Acid concentrations (0.125 mg/ml) (G2 medium) in women undergoing single fresh and frozen blastocyst transfer.

DETAILED DESCRIPTION:
The single blastocyst-stage embryo transfer cycles will be randomised in a 1:1 allocation, with block sizes of 2 and 4 on the day of Embryo Transfer (ET). This randomisation process will be centrally managed via a web-based electronic data capture system and will be stratified according to the treatment center. The allocation sequence and the designated treatment will be completely concealed from the participating couples, clinicians - including those conducting the transfer procedures - and outcome assessors. Given the intrinsic viscous nature of EmbryoGlue, embryologists, who who are responsible for the procedures in the laboratory will not be subjected to blinding. Only at the end of the study, when data collection is completed, the allocation sequence will be revealed to the primary investigators.

ELIGIBILITY:
Inclusion Criteria:

1. All cycles with single blastocyst transfer will be considered eligible
2. Both fresh and cryopreserved embryo transfer cycles utilizing autologous oocytes
3. No age restriction will be applied
4. Informed consent was signed

Exclusion Criteria:

1. Uterine anatomic anomalies
2. Women with untreated hydrosalpines
3. Once couples have been enrolled in the trial, subsequent cycles will not be incorporated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 858 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Live birth is defined as the birth of at least one live baby after 24 weeks of gestation.
  The primary outcome was Live birth rate per embryo transfer.

SECONDARY OUTCOMES:
Biochemical pregnancy | 12 days after embryo transfer.
  Biochemical pregnancy is defined as serum beta-human chorionic gonadotropin β-hCG > 20 IU/L 12 days after embryo transfer.
Clinical pregnancy | 6-8 weeks after embryo transfer
  Clinical pregnancy is defined as the presence of at least one gestational sac confirmed by ultrasonography (ectopic pregnancy is included as a clinical pregnancy).
Ongoing pregnancy | after 12 weeks of gestation.
  Ongoing pregnancy is defined as the presence of a gestational sac and fetal heartbeat after 12 weeks of gestation.
Miscarriage | 20 weeks of gestation.
  Miscarriage is defined as spontaneous loss of an intrauterine pregnancy before 20 completed weeks of gestation.
Ectopic pregnancy | After 4 to 6 weeks of embryo transfer
  Ectopic pregnancy is defined as a pregnancy implanted outside the uterine cavity, diagnosed by ultrasonography, surgical visualization, or histopathology.
Multiple pregnancy | 7 weeks of gestation.
  Multiple pregnancy is defined as a pregnancy with two or more gestational sacs or fetal heartbeats at 7 weeks of gestation.
hypertensive disorders in pregnancy | From 20 weeks of gestation up to at birth
  Comprising essential hypertension; pregnancy induced hypertension; pre-eclampsia and eclampsia.
Placental implantation disorders | From 20 weeks of gestation up to at birth
  Placental implantation disorders encompass placenta previa, placenta accreta spectrum, placental abruption and/or abnormal cord insertion
Preterm birth | At birth
  Delivery of a fetus at less than 37 and more than 28 weeks gestational age
Preterm premature rupture of membranes | Before 37 weeks of gestation and before the onset of labor
  Preterm premature rupture of membranes is defined as the leakage of amniotic fluid through the cervical os before 37 weeks of gestation and before the onset of labor
Mode of delivery | At birth
  Vaginal delivery or cesarean delivery
Gestational age | At birth
  Gestational age recorded at delivery
Birth weight | At birth
  Weight of baby born (grams)
low birth weight | At birth
  Weight of baby born < 2500 g
Very low birth weight | At birth
  Weight of baby born < 1500 g
Mean birth weight | 1 year after embryo transfer
  By checking medical records
Macrosomia | At birth
  Weight of baby born > 4000 g
Large for gestational age | At birth
  Birthweight > 90th percentile
Small for gestational age | At birth
  Birthweight < 10th percentile
Neonatal intensive care unit admission | Birth up to 1 year
  Safety outcome. Number of pregnancies for which newborn is admitted to the NICU
Stillbirth or late fetal death | At birth
  Fetal death at 20 or more weeks' gestation
Early neonatal death | Up to 28 days after birth
Congenital anomaly or birth defect | Birth to first year of life
  Any congenital anomalies detected in baby born

CONTACTS AND LOCATIONS:
Overall Officials: Juanzi Shi, Doctor, Study Chair — Center for Reproductive Medicine, Northwest Women's and Children's Hospital, Xi'an, Shaanxi, China
Locations (1):
- IVF laboratory, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Cai H, Xu D, Wang Z, Huang B, Xue X, Bai H, Man Y, Lei D, Wu Q, Ni Y, Lei J, Shi J. Efficacy and safety of hyaluronic acid-enriched transfer medium in women undergoing single blastocyst transfer: a study protocol for a multicentre randomised controlled trial. BMJ Open. 2025 Nov 19;15(11):e104571. doi: 10.1136/bmjopen-2025-104571. PMID 41263844